CLINICAL TRIAL: NCT00909805
Title: Interest of 2-octyl-cyanoacrylate (Dermabond®) in Closing Surgical Incisions in Children Before Acquisition of Continence. Randomised, Prospective, Non-inferiority Study.
Brief Title: Interest of 2-octyl-cyanoacrylate (Dermabond®) in Closing Surgical Incisions in Children Before Acquisition of Continence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Fondation Lenval (Other); Centre Hospitalier Régional Universitaire Montpellier (Other); Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-PP-10
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-02

CONDITIONS: Inguinal Incisions
Keywords: dermabond glue; suture; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cutaneous suture with glue (Experimental): Inguinal surgical incision closing using Dermabond® glue instead of cutaneous suture with surjet
  Interventions: Device: 2-octyl-cyanoacrylate (Dermabond® glue)
- Conventional suture (Active Comparator): Inguinal surgical incision closing with conventional cutaneous suture (surjet)
  Interventions: Device: cutaneous suture (Surjet)

INTERVENTIONS:
Device: cutaneous suture (Surjet) — cutaneous surjet suture
  Arms: Conventional suture
Device: 2-octyl-cyanoacrylate (Dermabond® glue) — the cutaneous suture is made with glue only
  Other Names: 2-octyl-cyanoacrylate (Dermabond®)
  Arms: Cutaneous suture with glue

SUMMARY:
Inguinal incisions are the most frequent incisions used in children before the acquisition of continence (180 incisions per year for the Pediatric Surgery Department in Nice CHU). However, healing of those wounds can be made hard because of soiling induced by urine and/or stool, which is unavoidable in case of wearing nappies.

Nowadays, in order to overcome a possible contamination of the surgical wound, post-surgery wound dressing is protected by the application of a waterproof band aid (like Tegaderm®) during wound-healing (evaluated to a mean of 7 days). When the band aid is soiled, a nurse changes it, causing unpleasantness in low age children (whose epidermal fragility is well known), and sometimes parents worry.

Moreover, those occlusive wound dressings avoid any control of the surgical wound during healing phase.

At the end of the wound-healing time, wound dressings are removed, causing discomfort for children and necessity of a qualified nurse staff at visit times.

Cutaneous use glues, introduced in surgery more than 10 years ago, allow making waterproof and transparent sutures, with a firmness equivalent to a 2/0 string suture (cutaneous suture in children is made with 5/0) and has its own local antiseptic properties. It does not need to be covered by any wound dressing during wound-healing phase. Moreover, cosmetic results for the 2-octyl-cyanoacrylate in the adult and children series (without any precise age distinction) seem to be equivalent to conventional sutures. Finally, its application goes with time saving (in preoperative and during wound-healing phase) and increases comfort for patients.

The aim of this study is to evaluate the efficiency of cutaneous use glue Dermabond® (2-octyl-cyanoacrylate) in surgical inguinal incisions sutures in children before the acquisition of continence, by a non-inferiority randomized multicentric prospective study.

Two patient groups will be studied, the sutures of one control group will be made with a conventional technique (intradermic surjet surgical suture), and one patient group will be sutured with 2-octyl-cyanoacrylate. The principal evaluation criteria is the suture quality (short- and long-term cosmetic aspect) evaluated by the surgeon.

Two secondary criteria will be studied :

* Parental satisfaction
* Ease of clinical nursing management Each studied criteria will be evaluated by a numeric score.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 24 months old
* Continuous nappies wearing for non-acquisition of continence
* Need of a surgical intervention which entry way is an inguinal incision in the inguinal fold (POTTS incision) for the following indications:

  * inguinal hernia
  * testicular ectopy
  * hydrocele
  * chord cyst
* Surgical incision smaller than 5 cm
* Informed consent form signed by both parents or by the legal representative
* Patient affiliated to French national health and pensions organization

Exclusion Criteria:

* Chronic or acute dermatological affection that can hamper wound-healing (atopic pathology, infectious pathology…)
* General affection that can hamper wound-healing (chronic denutrition)
* Cutaneous infection at the incision site
* Scar in the concerned region
* Medical history of wound-healing trouble
* Digestive pathology causing chronic or acute diarrhea
* Allergy to one of the used compounds (glue, string, wound dressing)
* Operative indication set in emergency with immediate surgery
* Non-acceptance of the protocol, refusal to participate to the study by one of the parents or the legal representative
* Impossibility of doing the follow up of the child, in accordance with the pre-established rules of the protocol

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Adequate or suboptimal wound-healing rate defined by a HOLLANDER cosmetic score higher or equal to 5 at the end of the initial wound-healing period. | J7-J10 and J+ 6 month

SECONDARY OUTCOMES:
Re-evaluation of the HOLLANDER cosmetic score 6 month after wound-healing. | J0, J7-J10 and J + 6 month
Parental satisfaction: 0-100 numeric scale divided in 5 items. | J0, J7-J10 and J + 6 month
Nurse satisfaction : 0-100 numeric scale divided in 4 items. | J0, J7-J10 and J + 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean BREAUD, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (4):
- France (4):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet2, Nice, Alpes Maritimes
  - Fondation Lenval -Hôpital Pédiatrique, Nice, Alpes Maritimes
  - Assistance Publique Hopitaux de Marseille - Hôpital Timone Enfants, Marseille, Bouches Du Rhône
  - Centre Hospitalier Universitaire de Montpellier - Hôpital Lapeyronie, Montpellier, Hérault